CLINICAL TRIAL: NCT00687726
Title: The Relationship of Knee Joint Osteoarthritis to Balance and Walking Ability.
Brief Title: Simple Home-Based Exercise for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Srinakharinwirot University (Other)
Responsible Party: Kanda Chaipinyo, Faculty of Health Science, Srinakharinwirot University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 056/2547
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2008-06-02 (Estimated); Status verified 2008-05

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; knee; exercise; balance
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- G1 (Experimental): Standing balance and mini squat training
  Interventions: Behavioral: Standing balance exercise
- G2 (Active Comparator): Isometric knee extension exercise
  Interventions: Behavioral: Isometric knee extension exercise

INTERVENTIONS:
Behavioral: Standing balance exercise — Standing balance and mini squat exercise performed 30 times/day/side, 5 days/week, for 4 weeks.
  Arms: G1
Behavioral: Isometric knee extension exercise — Isometric knee extension exercise performed 10 repetitions/set, 3 sets/day, 5 days/week for 4 weeks
  Arms: G2

SUMMARY:
1. Simple home-based standing balance training and isometric knee extension exercise for 4 weeks would improve functional ability and knee muscle strength of patients with knee osteoarthritis.
2. The outcome of standing balance training is different from isometric knee extension exercise.

ELIGIBILITY:
Inclusion Criteria:

* Clinical criteria for knee osteoarthritis

Exclusion Criteria:

* cardiovascular disease
* Parkinsonism
* osteoporosis
* inability to walk for 15 meters
* intra-articular injections

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-05; Primary Completion 2007-08 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Knee osteoarthritis outcome scores (KOOS) | 4 weeks

SECONDARY OUTCOMES:
Knee muscle peak torque | 4 weeks
Aggregate functional performance time | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kanda Chaipinyo, PT,PhD., Principal Investigator — Srinakharinwirot University
Locations (1):
- Faculty of Health Science, Srinakharinwirot University, Ongkharak, Changwat Nakhon Nayok, Thailand

REFERENCES:
- [Derived] Chaipinyo K, Karoonsupcharoen O. No difference between home-based strength training and home-based balance training on pain in patients with knee osteoarthritis: a randomised trial. Aust J Physiother. 2009;55(1):25-30. doi: 10.1016/s0004-9514(09)70057-1. PMID 19226239